CLINICAL TRIAL: NCT00704483
Title: A 12-week, Open Label, Multicenter, Titration Study, With a 9-month Maintenance Treatment Extension, to Demonstrate Efficacy of SBR759 Compared to Sevelamer HCl in Lowering Serum Phosphate Levels in Chronic Kidney Disease Patients on Hemodialysis
Brief Title: Efficacy of SBR759 in Lowering Serum Phosphate Levels in Chronic Kidney Disease Patients on Hemodialysis
Acronym: SBR759
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSBR759A2201; EUDRACT No.: 2006-001787-23
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2016-11

CONDITIONS: Hyperphosphatemia Patients With Chronic Kidney Disease on 3x/Week Replacement Therapy
Keywords: Chronic Kidney Disease; hemodialysis; hyperphosphatemia; hemodiafiltration
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperphosphatemia | interventions — SBR 759; Sevelamer

ARMS (4):
- 1 (Experimental): 1g tid
  Interventions: Drug: SBR759
- 2 (Active Comparator): Sevelamer HCl
  Interventions: Drug: Sevelamer HCl
- 3 (Experimental): SBR759 1.5 g tid
  Interventions: Drug: SBR759
- 4 (Active Comparator): Sevelamer HCl
  Interventions: Drug: Sevelamer HCl

INTERVENTIONS:
Drug: SBR759 — Starting dose of 1g or 1.5g tid, with an increase of 1g tid every 2 weeks until serum phosphate level fall below target.
  Arms: 1
Drug: Sevelamer HCl — 0.8 g tid
  Arms: 2
Drug: SBR759 — 1.5 g tid
  Arms: 3
Drug: Sevelamer HCl — 1.6 g tid
  Arms: 4

SUMMARY:
This study will evaluate the efficacy of SBR759 compared to sevelamer HCl in lowering serum phosphate levels in Chronic Kidney Disease patients on hemodialysis

ELIGIBILITY:
Inclusion criteria

* Men or women of at least 18 years old.
* Stable maintenance of renal replacement therapy 3 times per week.
* Controlled Serum phosphate if under phosphate-binder therapy.
* Serum phosphate level ≥ 6.0 mg/dL (> 1.9 mmol/L) prior to study treatment initiation.

Exclusion criteria

* Peritoneal dialysis.
* Parathyroidectomy or transplant scheduled during the study.
* Uncontrolled hyperparathyroidism
* History of hemochromatosis or ferritin > 1000 µg/L.
* Clinically significant GI disorder
* Unstable medical condition other than Chronic Kidney Disease.
* Treated with oral iron.
* Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2008-07; Primary Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Responder rates in target serum phosphate levels at 12 weeks Evaluate efficacy of SBR759 compared to sevelamer HCl at 12 weeks | Time Frame: 12 weeks + 12 months

SECONDARY OUTCOMES:
Responder rates in target patients with serum calcium-phosphate levels at 12 weeks/12 months | Time Frame: 12 weeks / 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (66):
- United States (19):
  - Novartis, Chula Vista, California
  - Novartis, La Mesa, California
  - Novartis, Whittier, California
  - Novartis, Denver, Colorado
  - Novartis, North Chicago, Illinois
  - Novartis, Peoria, Illinois
  - Novartis, Mishawaka, Indiana
  - Novartis, Baltimore, Maryland
  - Novartis, Fall River, Massachusetts
  - Novartis, Springfield, Massachusetts
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis, New York, New York
  - Novartis, Winston-Salem, North Carolina
  - Novarits, Fargo, North Dakota
  - Novartis, Portland, Oregon
  - Novartis, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Houston, Texas
  - Novartis, San Antonio, Texas
  - Novartis, Fairfax, Virginia
- Australia (6):
  - Novartis, Adelaide, South Australia
  - Novartis, Fitzroy, Victoria
  - Novartis, Parkville, Victoria
  - Novartis, Melbourne
  - Novartis, South Brisbane
  - Novartis, Woolloongabba
- Belgium (5):
  - Novartis Investigative Site, Antwerp
  - Novartis, Bruges
  - Novartis, Brussels
  - Novartis, Liège
  - Novartis Investigative Site, Saint Niklaas
- Canada (4):
  - Novartis Investigative Site, Edmonton
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Oshawa
  - Novartis Investigative Site, Québec
- Finland (4):
  - Novartis, Helsinki
  - Novartis, Oulu
  - Novartis, Tampere
  - Novartis, Turku
- France (5):
  - Novartis, Amiens
  - Novartis, Fleury-Mérogis
  - Novartis, Lyon
  - Novartis, Reims
  - Novartis, Salouël
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Coburg
- Italy (5):
  - Novartis Investigative Site, Lecco
  - Novartis Investigative Site, Lodi
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Modena
  - Novartis Investigative Site, Pavia
- Norway (4):
  - Novartis, Bergen
  - Novartis, Kristiansand
  - Novartis, Oslo
  - Novartis, Tønsberg
- Novartis, San Juan, Puerto Rico
- Sweden (4):
  - Novartis Investigative Site, Jönköping
  - Novartis Investigative Site, Karlstad
  - Novartis Investigative Site, Skövde
  - Novartis Investigative Site, Stockholm
- Switzerland (3):
  - Novartis, Aarau
  - Novartis, Lausanne
  - Novartis, Zurich
- United Kingdom (4):
  - Novartis, Hull
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Portsmouth
  - Novartis, Salford

REFERENCES:
- [Result] Chen JB, Chiang SS, Chen HC, Obayashi S, Nagasawa M, Hexham JM, Balfour A, Junge G, Akiba T, Fukagawa M. Efficacy and safety of SBR759, a novel calcium-free, iron(III)-based phosphate binder, in Asian patients undergoing hemodialysis: A 12-week, randomized, open-label, dose-titration study versus sevelamer hydrochloride. Nephrology (Carlton). 2011 Nov;16(8):743-50. doi: 10.1111/j.1440-1797.2011.01509.x. PMID 21854503
- See also: Results for CSBR759A2201 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=4645